CLINICAL TRIAL: NCT05743322
Title: The Usefulness of Pre-procedural 3D Print of Both Atria to Plan Transseptal Puncture for the Left Atrial
Brief Title: The Usefulness of Biatrial 3D Printing to Plan Transseptal Puncture for the Left Atrial Appendage Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Brno University Hospital (Other); General Teaching Hospital, Prague (Other)
Responsible Party: Principal Investigator, Pavel Osmancik, head of the dept. of cardiac arrhythmias, Charles University and University Hospital Kralovske Vinohrady, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3D PRINT FOR TSP
Record Dates: First submitted 2023-02-01; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Closure
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D printing arm (Experimental): A bi-atrial 3D printed model will be manufactured before the procedure
  Interventions: Device: Left atrial appendage closure

INTERVENTIONS:
Device: Left atrial appendage closure — Left atrial appendage will be occluded using commercially available device

SUMMARY:
The aim of the study is to assess the usefulness of pre-procedural 3D printing of both atria to plan optimum site for transseptal puncture for the left atrial appendage closure.

DETAILED DESCRIPTION:
All patients referred for the left atrial appendage closure will be enrolled. Before the procedure, cardiac CT (computed tomography) will be done. Using cardiac CT, segmentation procedure will be performed. The segmented 3D biatrial reconstruction will be exported in the stereolithography (STL) format and then printed out.

Before every procedure as a part of pre-procedural planning, TSP puncture will be simulated in vitro using the three-dimensional printing (3DP) models and a 12 Fr delivery sheath. Six holes (TSP locations) through the intraatrial septum will be performed from the right side of the septum by a cordless drill. The puncture sites will be localised as follows: three in the cranial part of the fossa ovalis (FO) (anteriorly just behind the aortic root, in the middle and posteriorly) and three in the caudal portion of the FO in the identical way. The delivery sheath will be inserted through each preformed hole and its distal tip was positioned in the LAA (10 - 20 mm deep). The relationship of the sheath and the proximal LAA segment will be evaluated in two orthogonal views. Two criteria had to be met in both views to classify the puncture site as optimal: (1) a central sheath position and (2) a coaxial sheath position (the angle with the LAA ostium axis not exceeding 30°).

All procedures will be done by experienced operators according to the actual guidelines. Intracardiac echocardiography (ICE) or transesophageal echocardiography (TEE) will be used. Before the procedure, each operator received a recommendation regarding the optimal puncture sites. In ICE guided cases, based on the LA anatomical structures visible in the projection plane during TSP, the puncture site was classified as posterior (left-sided pulmonary veins visible), middle (coumadin ridge visible), or anterior (LAA and mitral annulus visible). In TEE guided procedures mainly mid-oesophageal aortic valve short axis view (∼ 25-45°) and mid-oesophageal bicaval view (∼ 90-110°) will be used. Depending on in which third of the interatrial septum the puncture was performed, it will be classified as anterior, middle, or posterior (aortic valve short axis view). The bicaval projection showed the cranio-caudal localization.

The 3DP models were not used for device sizing, it was done based on the CT data and intra-procedural angiography according to the performing physicians' preferences.

The procedural difficulty will be assessed by the operator (focused on the alignment of the delivery assembly with the LAA axis). Furthermore, the number of recaptures of devices will be analyzed, as well as the number of unsuccessful procedures and procedural complications. Additional golas of the project are: to analyse the distribution of optimal puncture sites and to correlate CT 2D measurements with those findings.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation (paroxysmal or non-paroxysmal)
* CHA2DS2VASc more or equal 2 (Congestive heart failure, Hypertension, Age > 75 years, Diabetes, Stroke, Vascular disease, Age > 65 years, female sex)
* Contraindications for long-term anticoagulation

Exclusion Criteria:

* allergy to contrast dye
* non-willingness to participate
* left atrial appendage thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure satisfaction, scale 1-3 (1- optimum, 2-possible to implant, 3-impossible to implant) | It will be assessed immediately after the procedure, i.e. on the day of the procedure
  The satisfaction with the transseptal puncture for the purpose of the procedure, assessed by the operator
Angle between the delivery sheath and the LAA axis | It will be assessed immediately after the procedure, i.e. on the day of the procedure
  the axis between the delivery sheath with the axis of the left atrial appendage will be analysed in two orthogonal projections
Number of recaptures of the device | It will be assessed immediately after the procedure, i.e. on the day of the procedure
  Number of recaptures of the device

SECONDARY OUTCOMES:
Procedural complications | Until 30 days after the procedure
  Tamponade, device embolization, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Osmancik, Principal Investigator — Cardiac center University Hospital Kralovske Vinohrady
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared and available after the publication
Supporting Information: Study Protocol, CSR
Time Frame: After 6 months after the publication, on request
Access Criteria: On request